CLINICAL TRIAL: NCT02332356
Title: Therapeutic Optimization Study Based on MR Enterocolonography in Patients With Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Principal Investigator, Toshimitsu Fujii, MD PhD, Gastroenterology and Hepatology, Tokyo Medical and Dental University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MREC study
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Inflammatory Bowel Diseases; Disease Attributes
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Disease Attributes | interventions — Azathioprine; Adalimumab; Infliximab

ARMS (4):
- step up (Active Comparator): Procedure: MREC patients receive therapeutic step up
  Interventions: Drug: azathioprine or adalimumab and infliximab
- observation step up (No Intervention)
- step down (Active Comparator): Procedure: MREC patients receive therapeutic step down
  Interventions: Drug: azathioprine or adalimumab and infliximab
- observation step down (No Intervention)

INTERVENTIONS:
Drug: azathioprine or adalimumab and infliximab
  Arms: step down; step up

SUMMARY:
This randomized, controlled study aims to evaluate the impact of therapeutic intervention (step up) for the patients who are clinical remission with Magnetic Resonance Enterocolonography (MREC) active. In addition, to evaluate the impact of therapeutic step down for the patients who archived clinical and MREC remission. The primary endpoint is the rate of clinical remission at 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's and proven history of disease with clinical remission (CDAI<150)
* Signed written consent form to enroll the study (Need agreement from deputy for patients under 20years old)

Exclusion Criteria:

* Contraindication for infliximab, adalimumab, or azathioprine
* Lactating woman
* Presence of malignancy
* Within 3 month from intestinal surgery
* Presence of an end stoma
* Planned surgery

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The rate of clinical remission at 104 weeks. | 104 weeks

SECONDARY OUTCOMES:
The rate of hospitalization and operation | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Fujii, Principal Investigator — Tokyo Medical and Dental University Hospital
Locations (1):
- Gastroenterology and Hepatology, Tokyo Medical and Dental UNIV, Tokyo, Japan

REFERENCES:
- [Background] Takenaka K, Ohtsuka K, Kitazume Y, Nagahori M, Fujii T, Saito E, Naganuma M, Araki A, Watanabe M. Comparison of magnetic resonance and balloon enteroscopic examination of the small intestine in patients with Crohn's disease. Gastroenterology. 2014 Aug;147(2):334-342.e3. doi: 10.1053/j.gastro.2014.04.008. Epub 2014 Apr 13. PMID 24732015
- [Background] Hyun SB, Kitazume Y, Nagahori M, Toriihara A, Fujii T, Tsuchiya K, Suzuki S, Okada E, Araki A, Naganuma M, Watanabe M. Magnetic resonance enterocolonography is useful for simultaneous evaluation of small and large intestinal lesions in Crohn's disease. Inflamm Bowel Dis. 2011 May;17(5):1063-72. doi: 10.1002/ibd.21510. Epub 2010 Oct 25. PMID 21484957